CLINICAL TRIAL: NCT06931496
Title: Evaluation of the PROSTia Test in Patients Undergoing Prostate Biopsy
Acronym: PROSTIA- BP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, ESCHWEGE Pascal, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A02305-42
Record Dates: First submitted 2025-04-08; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: prostate cancer; risk calculator; Artificial intelligence
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prostia test (Experimental): patients who responded to the PROSTia questionnaire
  Interventions: Other: PROSTia test

INTERVENTIONS:
Other: PROSTia test — questionnaire with 50 questions

SUMMARY:
The investigators are interested here in the contribution of a new prostate cancer screening method and, more specifically, in the new and somewhat futuristic approach of artificial intelligence in the development of new, more accurate algorithms that make it possible to rethink the benefits of mass generalisation of prostate biopsies.

Main objective The main objective of this research is to use artificial intelligence and an associated algorithm to identify new indicators that would make it possible to avoid a prostate biopsy in patients with an initial suspicion of prostate cancer.

DETAILED DESCRIPTION:
.1. Outline of the study The lack of accuracy of the PSA test for prostate cancer screening leads to negative biopsies. The aim of this study is to determine whether the PROSTia test, a personalised medicine test using artificial intelligence (AI) by combining PSA, digital rectal examination (DRE) and 60 other qualitative data, could reduce the number of unnecessary biopsies and to estimate its impact on the detection of clinically significant cancers.

PROSTia employs the Gradient Boosting technique to select the variables of interest and optimise model performance. This process entails the utilisation of successive decision trees to model the non-linear relationships between the input variables and cancer risk. The construction of each tree is predicated on the correction of errors identified in preceding trees, with a focus on cases that have been misclassified. This iterative process is instrumental in generating a robust and accurate model for the purpose of prostate cancer screening

2 Methodology

The result of the PROSTia test is a score on a scale of 0 to 2. A score greater than or equal to 1 is considered a positive result. A positive result means that the patient has a significant risk of developing prostate cancer in the next 12 years. The following statistical analyses are performed using a 95% confidence interval:

* Sensitivity
* Specificity
* Positive likelihood ratio
* Negative likelihood ratio
* Disease prevalence
* Positive predictive value
* Negative predictive value
* Accuracy

Sensitivity, specificity, disease prevalence, positive and negative predictive values and accuracy are expressed as percentages.

Confidence intervals for sensitivity, specificity and accuracy are Clopper-Pearson 'exact' confidence intervals.

Confidence intervals for likelihood ratios are calculated using the logarithmic method as described on page 109 of Altman et al. 2000. Confidence intervals for predictive values are standard logit confidence intervals according to Mercaldo et al. 2007, except when the predictive value is 0 or 100%, in which case a Clopper-Pearson confidence interval is reported.

3. Number of patients The investigators set the number of patients at 150. This is a synthetic comparative study of a single patient cohort (i.e. there is no intervention as such; the cohort is compared to what it would be if the PROSTia test had been available).

Here are the assumptions that led to this number. Primary endpoint: binary (presence vs absence of disease).

Expected proportions: 50% in the study population (p2 without PROSTia) and 70% with PROSTia (p1).

Significance level (α): set at 0.05 Desired power (1-β): set at 0.8

Effect size: (p1-p2) drop rate:

The investigators plan to increase the calculated sample size to account for dropouts. calculated to account for dropouts or non-compliance with certain questionnaires (5%).

The method used to calculate the sample size is that of Woodward (1992).

4. Inclusion criteria

* Patients followed up at the Nancy CHRU in the Urology Department and eligible for prostate biopsy to screen for prostate cancer, taking into account an increase in PSA, PSA density,
* Adult males over 18 years of age
* Patients affiliated to or benefiting from a social security scheme
* Patients who understand French and are able to fill in a self-administered questionnaire or have someone to help them do so.

  5. Non-inclusion criteria
* Patient who has already undergone prostate biopsy
* Patient under court protection, guardianship or trusteeship
* Patient deprived of liberty by judicial or administrative decision

  6. Estimated time: Participation per person: Time taken to complete the questionnaire on the day of the biopsy of the biopsy (< 30 min) Duration of the inclusion period 12 months Total study duration 18 months

ELIGIBILITY:
Inclusion criteria:

* Patients followed up at the Nancy CHRU in the Urology Department and eligible for a prostate biopsy in search of prostate cancer, taking into account an increase in PSA, PSA density, lesion on MRI.
* Person who has received full information about the organisation of the research and has not objected to their participation and the use of their data.
* Adult male over 18 years of age - Patient affiliated to or benefiting from a social security scheme - Patient who understands French and is able to fill in a self-administered questionnaire or who has the possibility to be assisted in filling it in.

Exclusion criteria:

* Patients who have already had a prostate biopsy
* Patients under court protection, guardianship or trusteeship
* Patients deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity | Immediately after to notification of prostate biopsy results.
  Measuring the sensitivity of the test in comparison with the results of prostate biopsies
specificity | Immediately after to notification of prostate biopsy results.
  Measuring the specificity of the test in comparison with the results of prostate biopsies
positive likehood ratio | Immediately after to notification of prostate biopsy results.
  Measuring the positive likehood ratio of the test in comparison with the results of prostate biopsies
negative likehood ratio | Immediately after to notification of prostate biopsy results.
  Measuring the negative likehood ratio of the test in comparison with the results of prostate biopsies
disease prevalence | Immediately after to notification of prostate biopsy results.
  Measuring the disease prevalence of the test in comparison with the results of prostate biopsies
positive predictive value | Immediately after to notification of prostate biopsy results.
  Measuring the positive predictive value with the results of prostate biopsies
negative predictive value | Immediately after to notification of prostate biopsy results.
  Measuring the negative predictive value with the results of prostate biopsies
accuracy | Immediately after to notification of prostate biopsy results.
  Measuring the accuracy of the test in comparison with the results of prostate biopsies

SECONDARY OUTCOMES:
ability of the test to detect clinically significant cancers (ISUP ≥ 2) | Immediately after to notification of prostate biopsy results.
  Measuring the ability of the test to detect clinically significant cancers (ISUP ≥ 2) of the test in comparison with the results of prostate biopsies
failure rate of the test to detect the most aggressive cancers (ISUP 4 and 5) | Immediately after to notification of prostate biopsy results.
  Measuring the failure rate of the test to detect the most aggressive cancers (ISUP 4 and 5) of the test in comparison with the results of prostate biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France, France

IPD SHARING:
Plan to Share IPD: Undecided